CLINICAL TRIAL: NCT02411266
Title: Remote Ischemic Preconditioning to Ameliorate Delayed Ischemic Neurological Deficit After Aneurysmal Subarachnoid Hemorrhage: a Safety and Feasibility Study
Brief Title: Preconditioning With Limb Ischemia for Subarachnoid Hemorrhage
Acronym: PreLIMBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sebastian Koch, Associate Professor of Clinical Neurology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008 0406 II
Record Dates: First submitted 2015-03-30; First posted 2015-04-08 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): Subjects in this group will undergo sham preconditioning. A blood pressure cuff will be placed around the leg and inflated just lightly to a pressure of 30mmHg, not enough to affect arterial circulation. This will be maintained for 10min followed by 5min of deflation. This will constitute one conditioning cycle. There will be 3 sham conditioning cycles per treatment session.
  Interventions: Other: ischemic conditioning group
- treatment group (Active Comparator): Study personnel will place a blood pressure cuff around the subject's leg and use it to interrupt the circulation to the leg for 10 minutes followed by release of the blood pressure for 5 minutes. This will be repeated for a total of 3 times every 24 to 48 hours up to 14 days. The cuff will be inflated for 10 minutes and then deflated for 5 minutes. There will be 3 cycles of this. The cuff will be inflated to 200mmHg to induce ischemia, confirmed by palpation of pedal pulses.
  Interventions: Other: ischemic conditioning group

INTERVENTIONS:
Other: ischemic conditioning group — application of a blood pressure cuff around a leg and inflating the cuff to 200mmHg to induce limb ischemia for 10min followed by 5min reperfusion. this will be done for 3 cycles every 24-48hours during the first 14 days after subarachnoid hemorrhage
  Other Names: limb preconditioning

SUMMARY:
The purpose of this study is to learn about protecting the brain from dangerous low blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aneurysmal subarachnoid hemorrhage whose initial angiogram show an aneurysm and patients with clipped aneurysm will be eligible for enrollment.
* Patients will be enrolled within 96 hours of bleeding onset, if informed consent is obtained from the participant or health care proxy, as appropriate.

Exclusion Criteria:

* Hunt Hess Scale > 4
* Inability to undergo limb preconditioning due to local wound or tissue breakdown, history of peripheral extremity vascular disease or patient discomfort.
* Inability to obtain informed consent from the patient or a health care proxy.
* Ankle-brachial index < 0.7
* Inability to start limb preconditioning within 4 days of bleeding.
* Inability to precondition a leg that is not-plegic (that is preserved anti- gravity strength) and has not been accessed for catheter angiography
* Age<18 years
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-07-30 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Safety Outcomes 1 - number of patients who develop deep vein thrombosis and thromboembolism | 90 days
  The number of patients who develop deep vein thrombosis and thromboembolism in the treatment and control group.
Safety Outcome 2 - number of patients who develop neurovascular injury | 90 days
  The number of patients who develop neurovascular injury in the treatment and control group.
Safety Outcome 3 - number of patients who cannot tolerate the intervention due to discomfort | 90 days
  The number of patients who cannot tolerate the intervention due to discomfort.
Safety Outcome 4 - number of patients with cardiovascular events | 90 days
  The number of patients with cardiovascular events [defined as hypotension, myocardial ischemia]

OTHER OUTCOMES:
Clinical Outcome - number of patients with a good modified Rankin Scale, defined as less than 2 | 90 days
  The number of patients with a good modified Rankin Scale, defined as less than 2, in the control and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Koch, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No